CLINICAL TRIAL: NCT05013788
Title: Using Social Media to Decrease Healthcare Utilization for Pediatric Asthma: a Pilot Randomized Control Trial
Brief Title: Using Social Media to Decrease Healthcare Utilization for Pediatric Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Monica Kodakandla, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSC-MS-21-0426; UL1TR003167 (NIH)
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Asthma in Children
Keywords: Social Media; Pediatric Asthma; Healthcare Utilization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Other: Social Media Enhanced Education
- Control Group (Active Comparator)
  Interventions: Other: Usual Asthma Education

INTERVENTIONS:
Other: Social Media Enhanced Education — Along with usual asthma education received,participants will receive asthma education via various social media platforms ,Facebook, Twitter, Instagram, and/or Snapchat. Topics of education will include background on asthma and pathophysiology, asthma severity classification, asthma triggers, different medications and indications for when to take them, how to use an inhaler technique, and symptom monitoring.Online resources from the American Lung Association and the National Asthma Education and Prevention Program will also be posted.
  Arms: Treatment
Other: Usual Asthma Education — For patients who are admitted to Children's Memorial Hermann for asthma exacerbation, asthma education is provided to patients and families on the day of discharge by the nurse and respiratory therapist on triggers, Signs & Symptoms, Medication Use, Medication Delivery, Peak Flow, Zones and how to respond to each, and Cleaning equipment.Nursing staff are responsible for printing out education sheets to give to patients and showing an education video that is 20 minutes long. An asthma action plan are given to families on discharge. Patients that are discharged from the emergency room are given the same educational materials by the nurses and/or respiratory therapists except for the asthma video. Patients receive a variable amount of asthma education when going to usual clinic visits. The education provided is dependent on the provider, and usually limited in length to the time of the visit
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate if social media enhanced education (SME) will reduce total number of treatment days defined as summation of days of subsequent hospital admission, emergency room visits, and clinic visits, reduce missed school days, reduce total costs from a health system perspective, have increased effect with increased social media engagement, have increased effect in participants with both caregiver and patient (combined) with social media accounts, compared to participants where only the patient or only the caregiver uses social media (single),have increased patient satisfaction in the asthma education received and to obtain the experience and data needed to refine SME to be able to expand this platform for other chronic medical conditions with high healthcare utilization including pediatric diabetes, epilepsy, and sickle cell disease in children with asthma.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized to Children's Memorial Hermann admitted for asthma exacerbation
* patient and/or primary caregiver must have internet access on cellular phones or at home and use a social media account (Facebook, Twitter, Instagram, and/or Snapchat)

Exclusion Criteria:

* other chronic conditions besides asthma that may necessitate frequent health care utilization. i.e. children with complex chronic conditions, sickle cell, seizures, diabetes.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Kodakandla, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control Group
Started | 104 | 96
Completed | 102 | 95
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control Group | Total
Number analyzed (Participants) | 104 | 96 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.33 (3.57) | 7.29 (3.84) | 7.31 (3.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 48 | 102
  Male | 50 | 48 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 12 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 56 | 49 | 105
  White | 22 | 17 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 18 | 39
Region of Enrollment [Number; unit: participants]
  United States | 104 | 96 | 200

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Treatment Days in a Medical Setting (Hospital, Emergency Department (ED), Clinic)
Description: Treatment days are defined as the summation of days in the hospital, ED, or in the clinic.
Time Frame: 1 year after enrollment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 104 | 95
days | 1.97 (2.82) | 2.67 (5.18)

2. Secondary Outcome: Number of Days Hospitalized
Time Frame: 1 year after enrollment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 104 | 95
days | 0.12 (0.35) | 0.23 (0.61)

3. Secondary Outcome: Number of Participants With Hospital Readmissions
Time Frame: 1 year after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 104 | 95
Participants | 11 | 16

4. Secondary Outcome: Number of Participants With Emergency Room Visits
Time Frame: 1 year after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 104 | 95
Participants | 28 | 35

5. Secondary Outcome: Total Number of Clinic Visits
Time Frame: 1 year after enrollment
Measure: Mean (Standard Deviation); unit: clinic visits
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 104 | 95
clinic visits | 1.13 (1.78) | 1.17 (2.1)

6. Secondary Outcome: Patient Satisfaction and Understanding of Asthma Education
Description: This outcome was assessed using a questionnaire item asking, "How satisfied are you with the amount of asthma education provided to you?" The question is scored from 1 to 5, a higher number indicating a better outcome.
Time Frame: 1 year after enrollment
Population: Data were only collected for the participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 48 | 38
score on a scale | 4.71 (0.5) | 3.95 (1.07)

7. Secondary Outcome: Number of Missed Days of School
Time Frame: 1 year after enrollment
Population: Data were only collected for the participants who completed the survey.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 49 | 39
days | 3.8 (4.68) | 7.03 (10.25)

8. Secondary Outcome: Total Estimated Health System Costs, Hospital Costs, and Clinic Costs
Time Frame: 1 year after enrollment
Population: Data were not collected or analyzed for this outcome because cost data could not be obtained from the hospital and no cost information was available for participants. The study protocol was not amended to reflect this collective team decision. Data collection and analysis for this outcome measure will not be conducted in the future. Therefore, no participants were measured or analyzed for this outcome measure.
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 1 year after enrollment
Arm/Group | Treatment | Control Group
All-Cause Mortality (participants affected / at risk) | 0/104 | 1/96
Serious Adverse Events (participants affected / at risk) | 11/104 | 16/96
Other Adverse Events (participants affected / at risk) | 0/104 | 0/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=104) | Control Group (N=96)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 11 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT05013788/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT05013788/ICF_001.pdf